CLINICAL TRIAL: NCT03889600
Title: Addressing Social Determinants in Diabetes Care: The REDD-CAT Health-related Social Needs Screening Tool
Brief Title: Re-Engineered Discharge for Diabetes-Computer Adaptive Testing (REDD-CAT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was never conducted due to Covid. Key informant interviews were conducted instead.
Sponsor: Boston Medical Center (Other)
Collaborators: University of Michigan (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H-38545; R21DK121092 (NIH)
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Social determinants; Readmission
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REDD-CAT Recipient (Experimental): The nurse care manager will incorporate the administration of the REDD-CAT to the patient as part of the standard care discharge planning. He or she will utilize the REDD-CAT results report as a guideline for generating appropriate referrals to address unmet social needs identified.
  Interventions: Other: REDD-CAT

INTERVENTIONS:
Other: REDD-CAT — After obtaining informed consent from a participant and gathering baseline data, the study RA will send a flag in the EMR to notify the nurse care manager that a patient has enrolled in the REDD-CAT pilot. The nurse care manager will then incorporate the administration of the REDD-CAT to the patient as part of standard care discharge planning. He or she will utilize the REDD-CAT results report as a guideline for generating appropriate referrals to address unmet social needs identified.

SUMMARY:
Over 27 million Americans are diagnosed with Type 2 Diabetes Mellitus (T2DM), and their health outcomes, including hospitalization, emergency department use, and hospital readmission, are largely driven by social determinants; diabetes complications are largely attributable to unmet health-related social needs. Investigators will conduct a pilot feasibility trial of the Re-Engineered Discharge for Diabetes-Computer Adaptive Testing (REDD-CAT) system to inform the design of a future, fully-powered randomized controlled trial. REDD-CAT will allow clinical staff to preemptively link patients with community-based social services tailored to meet their unique needs in order to reduce avoidable hospitalization and emergency department visits.

DETAILED DESCRIPTION:
Investigators will conduct a pilot study with 30 patients to evaluate the feasibility and limited efficacy of the REDD-CAT social service screening and referral intervention to inform the design of a fully-powered trial. The study will determine the feasibility of delivering the REDD-CAT intervention in a clinical, point-of-care context to inform the design and implementation strategy for a fully powered clinical trial. It is not the purpose of this pilot clinical trial to determine sample size for a larger, fully-powered trial, as investigators already have data from prior readmissions research supporting sample size and power estimates using readmission rates as a primary outcome measure. After obtaining informed consent from a participant and gathering baseline data, the study research assistant (RA) will send a flag in the electronic medical record (EMR) to notify the nurse care manager that a patient has enrolled in the REDD-CAT pilot. The nurse care manager will then incorporate the administration of the REDD-CAT to the patient as part of standard care discharge planning. He or she will utilize the REDD-CAT results report as a guideline for generating appropriate referrals to address unmet social needs identified. To inform secondary measure selection for a future larger study, the RA will administer to enrolled patients a number of standardized measures, including the PHQ-9, GAD-7, Ways of Coping Questionnaire, and Diabetes Distress Scale. All baseline measures will be re-administered at 30-day follow-up to patients via the telephone. Data on hospitalizations and ED visits during the 30-day period post-discharge will be obtained from patients' medical records, and all data gathered will be stored in a REDCap electronic database.

ELIGIBILITY:
Inclusion Criteria:

* Boston Medical Center inpatient
* Lives in the greater Boston area
* Diagnosis of Type 2 diabetes
* English- speaking
* Demonstrated willingness and capacity to consent
* Age 18 or older
* Has reliable telephone access

Exclusion Criteria:

* Currently pregnant
* Has plans to leave the area for >2 weeks in the 45 days following enrollment in the study
* Diagnosis of dementia, memory loss, or memory deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-02 (Estimated); Primary Completion 2021-04-13 (Estimated); Study Completion 2021-04-13 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment potential: percentage of eligible patients willing to enroll in the study | 6 months
  Recruitment potential will be measured according to the percentage of eligible patients willing to enroll in the study. The source of this outcome data will be the hospital census and recruitment data.
Feasibility - Participant burden: time required for participants to complete data collection measures | 6 months
  Participant burden will be measured according to the time required for participants to complete data collection measures; the data source will be data collected by research assistants
Feasibility - Subject retention: percentage of patients who complete the 30-day follow-up time point | 30 days
  Retention will be measured according to the percentage of patients who complete the 30-day follow-up time point; study records will provide this data.
Feasibility - Implementation fidelity: percentage of indicated referrals that are made | 30 days
  Implementation fidelity will be measured according to the percentage of indicated referrals that are made; discharge records and electronic medical records will provide this data.

SECONDARY OUTCOMES:
Limited Efficacy - Change in coping: Ways of Coping scale | baseline, 30 days
  Coping will be assessed using the Ways of Coping scale which is a 66 item scale with potential responses from 1 to 4, with higher scores indicative of more frequent use of a particular strategy.
Limited Efficacy - Change in diabetes related distress: Diabetes Distress scale | baseline, 30 days
  Diabetes related stress will be assessed using the Diabetes Distress scale which comprises 17 items with potential responses ranging from 1 to 6, with lower scores indicating that an item is less of a problem and higher scores indicating that an item poses a greater problem.
Limited Efficacy - Change in depression: Patient Health Questionnaire (PHQ-9) | baseline, 30 days
  Change in depression will be assessed using the Patient Health Questionnaire (PHQ-9), which is a 9-item questionnaire that asks how often an individual has been bothered by a given item over the last 2 weeks. Scores range from 0 ("not at all") to 3 ("nearly every day.") A higher overall score indicates a greater level of depression.
Limited Efficacy - Change in anxiety: The Generalized Anxiety Disorder 7 (GAD-7) | baseline, 30 days
  The Generalized Anxiety Disorder 7 (GAD-7) will be used to assess changes in anxiety. The GAD-7 is a 7-item questionnaire that asks how often an individual has been bothered by a given item over the last 2 weeks. Scores range from 0 ("not at all") to 3 ("nearly every day.") A higher overall score indicates a greater level of anxiety.
Limited Efficacy - 30-Day readmission rate | 30 days
  30-Day readmission rate will be measured according to the percent difference between readmission rates for a historical control versus pilot readmission rates; this data will be collected via the EMR and clinical data warehouse

OTHER OUTCOMES:
Process Outcome- Referral Completion: percentage of patients who receive services post-referral | 30 days
  Referral Completion will be measured by the percentage of patients who receive services post-referral

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne E Mitchell, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03889600/ICF_000.pdf